CLINICAL TRIAL: NCT01072578
Title: An Open-label, Randomised, Two-period Crossover Study to Assess the Effect of Dapagliflozin on Percent Inhibition of Glucose Re-absorption When Administered Once a Day (10 mg OD) Versus Twice a Day (5 mg BID) in Healthy Male and Female Volunteers
Brief Title: A Study to to Assess the Effect of Dapagliflozin When Administered Once a Day Versus Twice a Day on Blood Glucose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D1691C00004
Record Dates: First submitted 2010-02-19; First posted 2010-02-22 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Inhibition of glucose re-absorption; diabetes; dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dapagliflozin
- 2 (Experimental)
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin tablets 5 mg, Oral Twice daily dose for 5 days (total daily dose 10 mg)
Drug: Dapagliflozin — Dapagliflozin tablets, 10 mg, Oral, once daily dose for 5 days

SUMMARY:
The primary objective of the study is to assess the effect of dapagliflozin on the amount of glucose in the blood and urine when dapagliflozin is administered once a day (10 mg) versus twice a day (5 mg every 12 hours) after five days of dosing.

ELIGIBILITY:
Inclusion Criteria:

* Female healthy volunteers must be post-menopausal (cessation of menses >1year, be surgically sterile (documented) or have undergone hysterectomy) or be sexually abstinent from enrolment until follow-up examination
* Have normal physical exam, vital signs ECG findings, and laboratory values

Exclusion Criteria:

* Use of prescription medication for a chronic or acute medical condition within 3 weeks of randomization
* History or presence of neurological, haematological, psychiatric, gastrointestinal, hepatic or renal disease, or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs as determined by the Investigator
* Previous participation in an AstraZeneca (AZ) or Bristol-Myers Squibb (BMS) dapagliflozin study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Calculation of derivation of pharmacokinetic variables | Up to 14 blood samples will be obtained on day 1 (with the closest interval between samples being 15 minutes), one sample on days 3 and 4, and up to 21 samples on day 5

SECONDARY OUTCOMES:
Calculation of derivation of pharmacodynamic variables (inhibition of plasma glucose re-absorption, 24 hour urine glucose excretion, inhibition of rate of gut glucose absorption by measuring plasma glucose, insulin and GIP). | plasma glucose will be drawn on Day 5, creatinine will be drawn at pre-dose of Day 4 and of Day 5, glucose and insulin will be drawn on Day 5 , Day 5 for GIP, urine will be collected on Day 5 in 4-hour intervals
To examine the safety and tolerability of the combination of dapagliflozin and metformin | Adverse events and laboratory variables assessed throughout both 5-day treatment periods, and a follow-up visit 5-10 days later

CONTACTS AND LOCATIONS:
Overall Officials: Georg Golor, Principal Investigator — Parexel; Thomas Koernicke, Study Director — Parexel
Locations (1):
- Research Site, Berlin, Germany

REFERENCES:
- [Derived] Tang W, Reele S, Hamer-Maansson JE, Parikh S, de Bruin TW. Dapagliflozin twice daily or once daily: effect on pharmacokinetics and urinary glucose excretion in healthy subjects. Diabetes Obes Metab. 2015 Apr;17(4):423-5. doi: 10.1111/dom.12425. Epub 2015 Jan 12. PMID 25511685